CLINICAL TRIAL: NCT02269956
Title: Mealtime Symptoms in Dementia: Adaptive Leadership Approaches
Brief Title: Mealtime Symptoms in Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00055958
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Feasibility Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): The 2 NH's not used in the focus groups will receive the intervention, a 12-week feasibility study. At baseline, weeks 6 and 12, dementia feeding skills knowledge and self-efficacy tests will be administered, meal observations of nursing staff assisting PWD with meals will be video recorded for 3 meals over 2 days at baseline and again at week 6 and 12, and a medical record review will be conducted. After baseline data is collected, the training program will be delivered in 5 weekly modules with group coaching sessions completed the same week.
  Interventions: Behavioral: 12 week feasibility study
- Focus Groups (No Intervention): Year 1 focus groups will aim to identify how nursing staff feel about usual interventions for feeding behaviors of PWD and staff responses when a PWD displays difficult eating behaviors. Year 2 focus groups will evaluate the revised dementia feeding skills training program, the coaching interventions, and case scenarios, and indicate how realistic and compatible the intervention is with their work environment.

INTERVENTIONS:
Behavioral: 12 week feasibility study — : At baseline, weeks 6 and 12, dementia feeding skills knowledge and self-efficacy tests will be administered, meal observations of nursing staff assisting PWD with meals will be video recorded for three meals over two days, and a medical record review will be conducted to ascertain technical and adaptive interventions also in place for the PWD (e. g., high density protein supplements, appetite stimulant medications, weighing, diet texture modifications). After baseline data is collected, the training program will delivered in five weekly modules with group coaching sessions completed the same week
  Arms: Intervention

SUMMARY:
The purpose of this study is to combine current evidence-based guidelines with adaptive leadership (AL) training to assist nursing staff to navigate the delicate balance of necessary technical and adaptive work to improve problematic dementia-related mealtime symptoms.

DETAILED DESCRIPTION:
Currently, basic training programs do not adequately teach nursing home (NH) staff to handle behavioral symptoms at mealtime that typically accompany dementia. When persons with dementia (PWD) exhibit mealtime symptoms (e.g. turning away of the head, pushing food away), these symptoms may be interpreted as lack of interest in eating, and feeding attempts ceased. This misinterpretation poses serious health risks to PWD including under-nutrition and increased risk for more aggressive medical treatment (e.g. feeding tube). The Aims of this study are to: 1) Identify the adaptive leadership challenges of NH staff for alleviating mealtime symptoms for PWD; 2) Determine NH staff evaluation of a dementia feeding skills training program that combines adaptive leadership approaches with technical approaches to mealtime symptoms; and 3) Conduct a 12-week feasibility study implementing this dementia feeding skills training program with NH staff, linking training to resident outcomes. Focus groups will be conducted in four NHs during which NH staff will describe adaptive challenges around: mealtime symptom recognition, communication patterns, typical responses to mealtime symptoms, and feelings when interventions are met with success or failure. Focus group interviews will be transcribed and content analysis conducted. Findings from the focus group interviews will be used to revise a dementia feeding skills program. The revised training program will be evaluated by NH staff to determine how NH staff perceives the coaching intervention, and if case scenarios are realistic and compatible with current workplace practices. The training program will be implemented in two skilled NHs over a five week period. NH staff outcomes include mealtime knowledge and self-efficacy. Through meal observations, NH staff will be assessed for time spent assisting with feeding and feeding skill behaviors; and PWD outcomes assessed by quantifying meal intake and aversive feeding behaviors. Findings from this study will describe adaptive leadership challenges for NH staff, revise and implement a training program teaching NH staff adaptive and technical interventions for alleviating mealtime symptoms for PWD in the NH setting.

ELIGIBILITY:
Inclusion Criteria:

Nursing Home staff participants must be:

1. 18 years of age or older,
2. able to read and write English,
3. willing to sign informed consent,
4. employed as a Registered Nurse, Licensed Practical Nurse, Certified Nursing Assistant, part of the Nursing Home Administration team, or part of the therapy team.

Persons With Dementia participants must be:

1. a resident (> 6 wks) of NH,
2. 60+ years of age,
3. able to speak English in order to give assent,
4. have a positive Minimum Data Set 3.0 for: Active disease diagnosis of Alzheimer's Disease or dementia,
5. require extensive assistance to total dependence for eating,
6. have a Brief Interview for Mental Status (BIMS) score ranging from 0-12 (lower score indicates greater cognitive impairment)37, and
7. have a legally authorized representative (LAR) able to read English in order to provide informed consent for the PWD.

Exclusion Criteria:

PWD:

* Minimum Data Set 3.0 positive for: Human Immunodeficiency Virus (HIV) Infection, Parkinson's Disease, and/or Traumatic Brain Injury,
* any swallowing disorder,
* parental/ IV feedings, or presence of a feeding-tube;
* any significant auditory or visual impairment that would prevent the PWD from hearing/seeing verbal/visual cues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Feeding Skills Knowledge Test | Baseline (before training program), Week 6 (after training program), and Week 12
  10 item multiple choice test administered in paper/ pencil format to nursing staff assisting with feeding persons with dementia (Scores range from 0-10)
Change in Feeding Skills Self-Efficacy Test | Baseline (before training program), Week 6 (after training program), and Week 12
  10 items with likert scale response administered to nursing home staff

SECONDARY OUTCOMES:
Functional Rating Scale for Symptoms in Dementia | 12 weeks
  14 categories related to functional ability of PWD (e. g., eating and dressing ability, emotionality, memory). Each category scores 0-3. Totals range from 0-42; higher score indicative of greater impairment
Brief Inventory of Mental Status | 12 weeks
  Part of Minimum Data Set (MDS) 3.0. 5 sections of cognitive ability questions scored 0-2; scores of 0-12 considered moderate to severe cognitive impairment.
C3P Feeding Skills Checklist | 12 weeks
  Multi-item checklist of feeding skill behaviors grouped around changing the person, place or people. Each section is given numerical value.
Food Intake Record | Collected for 3 meals over 2 days at Baseline, Week 6 and Week 12
  Meal intake documented by pre-post meal tray weight as well as documentation of hand feeding techniques used during the meal.
Edinburgh Feeding in Dementia (EdFED) scale | Collected for 3 meals over 2 days at Baseline, Week 6 and Week 12
  Scale measuring aversive feeding behaviors on a 0-20 scale of 10 items. Higher scores equal more aversive feeding behaviors.
Time Spent Feeding | Collected for 3 meals over 2 days at Baseline, Week 6 and Week 12
  Time spent feeding was measured in hours and minutes via stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Batchelor-Murphy, PhD, Principal Investigator — Duke University School of Nursing

REFERENCES:
- [Derived] Liu W, Batchelor M, Williams K. Development and Psychometric Testing of the Mealtime Engagement Scale in Direct Care Providers of Nursing Home Residents With Dementia. Gerontologist. 2021 Nov 15;61(8):e410-e420. doi: 10.1093/geront/gnaa097. PMID 32726447
- [Derived] Liu W, Batchelor M. Mealtime Caregiving Engagement for Residents with Advanced Dementia: Item Response Theory Analysis. West J Nurs Res. 2021 Apr;43(4):374-380. doi: 10.1177/0193945920943898. Epub 2020 Jul 17. PMID 32680448